CLINICAL TRIAL: NCT01434433
Title: Alere Triage fs BNP Method Comparison Evaluation
Brief Title: Alere Triage fs B-type Natriuretic Peptide (BNP) Method Comparison Evaluation
Acronym: ABC
Status: Completed | Type: Observational
Sponsor: Alere San Diego (Industry)
Responsible Party: Sponsor
Organization: Abbott RDx Cardiometabolic (Other)
Other Study IDs: BSTE-9012
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Specimens With BNP Values of 5 to 5000 pg/ml; Triage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will evaluate method correlation and mean bias between six B-type natriuretic peptide (BNP) platforms.

ELIGIBILITY:
Inclusion Criteria:

* Samples with BNP range of 5-5000 pg/ml
* Samples with sufficient volume for testing

Exclusion Criteria:

* BNP <5 pg/ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department, Hospital
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
bias | Sept 2011

CONTACTS AND LOCATIONS:
Overall Officials: Fred Apple, M.D., Principal Investigator — Hennepin Healthcare Research Institute